CLINICAL TRIAL: NCT06776159
Title: The Effect of Standardizing Procedures for Subcutaneous Injections of Low-molecular-weight Heparin on Patients With Cardiovascular Diseases: A Cluster Randomized Controlled Trial
Brief Title: The Effect of Standardizing Procedures for SC Injections of LMWH on Patients With CVD
Acronym: LMWH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, CHEUNG Pui Yu Frankie, Assistant Professor of Practice, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20250301; CHEUNGPuiYu (Other: Hong Kong PolyU)
Record Dates: First submitted 2024-12-30; First posted 2025-01-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: CVD - Cardiovascular Disease; Bruise; Pain
Keywords: LMWH injection
MeSH Terms: conditions — Cardiovascular Diseases; Contusions; Pain

STUDY DESIGN:
Intervention Model Description: Double-blinded, two-armed, clustered randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The administrative staff, who will be responsible for data collection, will be masked for the group allocation during the whole process. The patients will be masked for the intervention purpose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control (Active Comparator): The control group participants will receive the usual practice of subcutaneous LMWH injection administered by nurses.
  Interventions: Other: Active Control
- Standardized injection protocol (Experimental): The intervention group participants will receive standardized LMWH injection administered by nurses.
  Interventions: Other: Standardized injection protocol

INTERVENTIONS:
Other: Active Control — Patients in the control group will receive the usual practice of subcutaneous LMWH injection administered by nurses.
  Arms: Active Control
Other: Standardized injection protocol — Nurses administer LMWH according to the standardized evidence-based protocol.
  Arms: Standardized injection protocol

SUMMARY:
Improper subcutaneous administration of LMWH may cause complications at the injection site. Standardized protocol for subcutaneous LMWH injections in patient with cardiovascular diseases is warranted to ensure consistent best practices in clinical settings.

DETAILED DESCRIPTION:
This study examines the effect of standardized protocol in reducing complications for patients with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* patients who are in cardiac care units suffering from cardiovascular diseases prescribed with LMWH injections two times per day
* Chinese

Exclusion Criteria:

* cognitively impaired
* unconscious
* refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Bruising | 24 hours, 48 hours, 72 hours
  The bruising diameter will be measured by a ruler and the incidence of bruising will be recorded.
Pain | Immediately after injection, 24 hours, 48 hours, 72 hours
  Patients' pain levels are assessed using the Verbal Descriptor Scale: 'severe pain,' 'moderate pain,' 'mild pain,' and 'no pain.' 'Severe pain' indicates the worst outcome, followed by 'moderate pain,' then 'mild pain,' with 'no pain' representing the best outcome.

SECONDARY OUTCOMES:
Patient Experience | Immediately after receiving the injection
  a Patient Experience Surveys to evaluate their perceived nurse's attitude
Communicative Competence | Immediately before and after injection
  Communicative Competence Scale consists of 36 items across five dimensions (General Competence, Empathy Affiliation/Support, Behavioural Flexibility, and Social Relaxation), using a 5-point Likert scales ranging from strongly agree to strongly disagree (coded from 1 to 5). Higher the score means worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hospital Authority, Hong Kong, Hong Kong, Hong Kong